CLINICAL TRIAL: NCT03174938
Title: The Swedish BioFINDER 2 Study
Acronym: BioFINDER2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Erik Stomrud, M.D., PhD, Skane University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BioFINDER 2
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Alzheimer Disease; Parkinson Disease; Lewy Body Disease; Parkinson-Dementia Syndrome; Frontotemporal Degeneration; Semantic Dementia; Progressive Nonfluent Aphasia; Progressive Supranuclear Palsy; Corticobasal Degeneration; Multiple System Atrophy; Mild Cognitive Impairment
Keywords: Early diagnosis, biomarker, PET, MRI, β-amyloid, tau, CSF, cognitive test
MeSH Terms: conditions — Dementia; Alzheimer Disease; Parkinson Disease; Lewy Body Disease; Progressive supranuclear palsy atypical; Frontotemporal Dementia; Primary Progressive Nonfluent Aphasia; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Multiple System Atrophy; Cognitive Dysfunction; Disease; Pick Disease of the Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- COHORT A: Cognitively healthy younger individuals (40-65 y) (Other): We will recruit 300 cognitively healthy individuals from the Malmö Offspring study, which is an epidemiological study. The participants will be stratified according to a) family history of dementia in first degree relatives (with onset before 80 years of age) and b) APOE 4 genotype; i.e. 25% will have no family history and no APOE4 allele, 25% will have a family history and no APOE 4 allele, 25% will have no family history and at least one APOE 4 allele, 25% will have a family history and at least one APOE 4 allele.
  FOLLOW-UP FOR 8 YEARS Every 2 years new clinical, cognitive, neurological, and psychiatric assessments will be performed as well as CSF/blood sampling.
  MRI, Tau PET and Amyloid PET will be done every 4 years in all cases, and Tau PET and MRI every two years if the subject is amyloid positive at baseline.
  An auxiliary cohort (termed "Cohort A2") of 40 healthy individuals aged 20-40 years of age will also be included.
  Interventions: Diagnostic Test: Flutemetamol F18 Injection; Diagnostic Test: [18F]-RO6958948; Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau; Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau
- COHORT B: Cognitively healthy elderly individuals (66-100 y) (Other): We will recruit 300 cognitively healthy individuals from the Malmö/Lund region, where we will aim to include as many individuals as possible that did participate in the Malmö Diet and Cancer study during the early 1990's. The participants will be stratified according to a) family history of dementia in first degree relatives (with onset before 80 years of age) and b) APOE 4 genotype; i.e. 25% will have no family history and no APOE 4 allele, 25% will have a family history and no APOE 4 allele, 25% will have no family history and at least one APOE 4 allele, 25% will have a family history and at least one APOE 4 allele.
  FOLLOW-UP FOR 8 YEARS Every 2 years new clinical, cognitive, neurological, and psychiatric assessments will be performed as well as CSF/blood sampling.
  MRI, Tau PET and Amyloid PET will be done every 4 years in all cases, and Tau PET and MRI every two years if the subject is amyloid positive at baseline. Motor assessments (Motor-ACT) are performed at baseline and afte
  Interventions: Diagnostic Test: Flutemetamol F18 Injection; Diagnostic Test: [18F]-RO6958948; Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau; Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau
- COHORT C: SCD and MCI (Other): >750 patients with either subjective cognitive decline (SCD) or mild cognitive impairment (MCI) will be recruited in a consecutive fashion from the Skåne University Hospital and Ängelholm Hospital. We will only include cases where the medical doctor believes that the cognitive symptoms are caused by an incipient neurocognitive disorder. For example, cases with evidence of brain amyloid pathology (i.e. an abnormal CSF Aβ42/40 ratio).
  FOLLOW-UP FOR 6 YEARS Every 12 months new clinical, cognitive, neurological, and psychiatric assessments will be performed.
  CSF/blood sampling, Tau PET, Amyloid PET and MRI will be done every 2 years. Motor assessment (Motor-ACT) at year 1, year 3 and year 5.
  A auxiliary cohort ("Cohort C2") >150 cases with SCD/MCI where the doctor does not suspect incipient neurocognitive disorder, will undergo the same baseline investigations, but they will be followed up clinically only after 2, 4 and 8 y.
  In total, 1000 patients with SCD or MCI will be included.
  Interventions: Diagnostic Test: Flutemetamol F18 Injection; Diagnostic Test: [18F]-RO6958948; Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau; Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau
- COHORT D: Dementia due to Alzheimer's disease (Other): 400 patients with mild to moderate dementia due to Alzheimer's disease (AD) will be recruited from the Skåne University Hospital and Ängelholm Hospital in southern Sweden. We will include at least 50 cases aged 40-65 years of age, at least 200 cases aged 66-79 years of age and at least 50 cases aged 80-100 years of age.
  FOLLOW-UP FOR 2 YEARS Every 12 months new clinical, cognitive, neurological, and psychiatric assessments will be performed.
  CSF/blood sampling, Tau PET and MRI will be done at baseline and after 2 years. Amyloid PET is performed at baseline for a subset of this group.
  Interventions: Diagnostic Test: [18F]-RO6958948; Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau; Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau
- COHORT E: Other dementias (Other): Patients with primary neurodegenerative disorders other than Alzheimer's disease will be recruited:
  1. 160 cases with Frontotemporal dementia (FTD)-related disorders, including behavioral variant of FTD (bvFTD), Progressive nonfluent aphasia (PNFA), semantic dementia (SD), Progressive supranuclear palsy (PSP), Corticobasal degeneration (CBD).
  2. 50 cases with subcortical Vascular dementia (VaD).
  3. 200 cases with either Parkinson's disease (PD), Parkinson's disease with dementia (PDD), Dementia with Lewy Bodies (DLB), Multiple system atrophy (MSA).
  FOLLOW-UP FOR 2 YEARS Every 12 months new clinical, cognitive, neurological, and psychiatric assessments will be performed.
  CSF/blood sampling, Tau PET (depends on further funding) and MRI will be done at baseline and after 2 years. No Amyloid PET in this group. Motor assessments (Motor-ACT) are performed at baseline and a 2-year follow-up since 7th Oct 2019.
  Interventions: Diagnostic Test: [18F]-RO6958948; Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau; Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau

INTERVENTIONS:
Diagnostic Test: Flutemetamol F18 Injection — PET imaging of Abeta amyloid
  Other Names: Vizamyl
  Arms: COHORT A: Cognitively healthy younger individuals (40-65 y); COHORT B: Cognitively healthy elderly individuals (66-100 y); COHORT C: SCD and MCI
Diagnostic Test: [18F]-RO6958948 — PET imaging of Tau aggregates
Diagnostic Test: Elecsys (Roche) Abeta42, Ttau and Ptau — Measurement of Abeta42, Ttau and Ptau in the cerebrospinal fluid
Diagnostic Test: Lumipulse (Fujirebio) Abeta42, Ttau and Ptau — Measurement of Abeta42, Ttau and Ptau in the cerebrospinal fluid

SUMMARY:
The Swedish BioFINDER 2 study is a new study that will launch in 2017 and extends the previous cohorts of BioFINDER 1 study (www.biofinder.se). BioFINDER 1 is used e.g. to characterize the role of beta-amyloid pathology in early diagnosis of Alzheimer's disease (AD) using amyloid-PET (18F-Flutemetamol) and Aβ analysis in cerebrospinal fluid samples. The BioFINDER 1 study has resulted in more than 40 publications during the last three years, many in high impact journals, and some the of the results have already had important implications for the diagnostic work-up patients with AD in the clinical routine practice.

The original BioFINDER 1 cohort started to include participants in 2008. Since then there has been a rapid development of biochemical and neuroimaging technologies which enable novel ways to the study biological processes involved in Alzheimer's disease in living people. There has also been a growing interest in the earliest stages of AD and other neurodegenerative diseases. With the advent of new tau-PET tracers there is now an opportunity to elucidate the role of tau pathology in the pathogenesis of AD and other tauopathies. The Swedish BioFINDER 2 study has been designed to complement the BioFINDER 1 study and to e.g. address issues regarding the role of tau pathology in different dementias and in preclinical stages of different dementia diseases. Further, the clinical assessments and MRI methods have been further optimized compared to BioFINDER 1. Detailed assessments of motor aspects and dual task performance, which is part of a sub-study named Motor-ACT: "Motor aspects and activities in relation to cognitive decline and brain pathologies, has been added to further optimize assessment of motor function.

DETAILED DESCRIPTION:
GENERAL AIMS:

1. Develop methods for early and accurate diagnosis of different dementia disorders. This is important not only for the clinical diagnostic work-up, but also for selection of patients to clinical trials. Because dementia is very common among the elderly, but often misdiagnosed, we need to develop minimally invasive, reliable and affordable biomarkers for use in a primary care setting. This could include blood-based biomarkers which could be used to identify patients at high risk for a neurodegenerative disease. We also aim to develop new diagnostic algorithms using advanced imaging techniques and cerebrospinal fluid (CSF) biomarkers to diagnose patients prior to overt symptoms (when brain dysfunction is still limited and potentially reversible) in order to identify individuals more likely to respond to new disease-modifying therapies.
2. Develop biomarkers and imaging techniques to monitor early effects of new disease-modifying therapies. Methods are needed that can reliably detect relevant changes in the turnover of Aβ, tau and α-synuclein. In the present study one focus will be to study the annual change in the retention of Tau PET ligands during both the prodromal and dementia stages of AD. Further, we need biomarkers that detect the intensity of ongoing synaptic/neuronal degeneration. Imaging methods revealing the functional and structural integrity of different brain networks might also be relevant.
3. Investigate the heterogeneity of dementia and parkinsonian disorders to assist in the development of a new pathology-based disease classification. Current diagnostic work-up is based on symptomatology. However, the diseases (e.g. Alzheimer's and Parkinson's diseases) are heterogeneous with respect to clinical features and underlying pathologies. Moreover, there is also significant overlap between the diseases. Hence, today's symptom-based clinical diagnostic criteria are likely too crude to provide an etiologically meaningful classification of patients. We will therefore work towards a pathology-based disease classification, using in vivo biomarkers that reflect the underlying brain pathologies, e.g. Aβ or tau. This will be especially useful for the development of new disease-modifying therapies, which are aimed at specific brain pathologies.
4. Define the temporal evolution of pathologies in the predementia phases of Alzheimer's disease. One of the last decade's paradigm shifts in neuroscience has been the realization that AD, and likely also other neurodegenerative diseases, starts with a prolonged predementia phase. AD even starts with an asymptomatic phase, when brain pathology is present in the absence of clinical symptoms. It has become clear that we need to better understand the temporal sequence of pathologic events in these disorders to be able to select the optimal disease stages for interventions in clinical trials with different disease-modifying therapies directed at specific pathologies.
5. Investigate the underlying disease mechanisms of dementia disorders in humans aiming at finding new relevant drug targets. Drug discovery using the currently available cell and animal models, has not translated to human research as indicated by failed phase II and III trials. There are several possible reasons for these failures. First, it is possible that previous trials may have focused on the wrong drug targets, since findings from cell and animal models of dementias may not have accurately captured essential aspects of the disease mechanisms in humans. BioFINDER2 will be a translational study where we will attempt to bridge the knowledge gap between cell/animal studies and studies in humans, by using biomarkers that reflect biological mechanisms that may be studied across model systems. Second, another reason of the failed trials may be that they included patients in too advanced disease stages for the treatments to be effective, or that they partly included patients with unspecific diseases, since they did not use biomarker-based methods for inclusion of participants. BioFINDER2 will inform on the design of future clinical trials by providing detailed data about cognitive and functional changes over time in people with well-defined biomarker-characterized brain pathologies.

STUDY PLAN To reach the objectives above, we include well-characterized and clinically relevant populations of patients with dementia and/or parkinsonian symptoms and healthy individuals. We apply several state of the art methodologies in order to develop new brain imaging techniques, new biomarkers in blood and CSF as well as novel methods of assessing important clinical symptoms.

COGNITIVE TESTING Attention and executive function will be assessed with the Trail Making Test A and B (TMT), Symbol Digit Modalities Test (SDMT), and A Quick Test of cognitive speed (AQT). Visuospatial ability will be measured by two subtests from the Visual Objects and Space Perception (VOSP) battery, incomplete letters and cube analysis. Memory will be assessed with the Free and Cued Selective Reminding Test (FCSRT) in cohorts A and B. It will be complemented with the 10-word delayed recall test from ADAS-cog, including a recognition part. Verbal ability will be evaluated with the animal and letter S fluency tests and the 15-item short version of the Boston Naming Test. Global cognition will be assessed with the Mini-Mental State Examination (MMSE). In cohort A and B, a computerized cognitive battery focusing on memory and attention will also be performed.

ASSESSMENTS OF SYMPTOMS, FUNCTIONAL ABILITIES AND GLOBAL FUNCTION Cognitive symptoms. All subjects will rate his or her memory and attention/executive function in relation to others of the same age according the Brief Anosognosia Scale (BAS). We have also added similar questions to cover the other cognitive domains. These questions have been validated against neuropsychological testing but there are data indicating that self-reported cognitive complaints are only valid in a lesser degree of cognitive impairment. To assess a broader range of cognitive complaints, the Subjective Cognitive Decline questionnaire (SCD-q) will be administered to the research subjects. Subjects from cohorts C, D and E will be assessed with cognitive impairment questionnaire (CIMP-QUEST; filled out by an informant).

Functional ability. This will be evaluated with the informant-based Functional Activities Questionnaire (FAQ) or the Amsterdam IADL scale, both focus on instrumental activities of daily living (IADL) known to be affected early in cognitive decline.

Global function. The global cognitive status will be evaluated using the sum of boxes score from the Clinical Dementia Rating scale (CDR) and the global deterioration scale (GDS).

Behavioral and psychological symptoms in dementia (BPSD). BPSD will be assessed by clinicians using the Neuropsychiatric Inventory - Clinician rating scale (NPI-C) developed by Jeffrey Cummings. Mood and anxiety will be further assessed with the Hospital Anxiety and Depression scale (HADS). Frontal Behavioral Inventory (FBI) will be done in FTD-related conditions.

Quality of Life (QoL). The overall health status will be rated by the subjects using the EQ-5D from Euro-QoL. In demented patients this will also be rated by an informant, spouse or close relative.

Sleep. The presence of REM sleep behavior disorder will be evaluated with a single validated composite question derived from the Mayo Sleep Questionnaire. Sleep quality is assessed with the Sleep Scale from the Medical Outcome Study (MOS).

Cognitive reserve. Premorbid cognition and cognitive reserve is approximated from the Cognitive Reserve Index questionnaire (CRI-q; subitems "Education" and "Working activity", not "Leisure time").

MOTOR ASSESSMENTS Motor aspects are evaluated as part of the sub-study Motor-ACT, which includes detailed motor assessments (including dual tasking): clinical assessments (administered by a physiotherapist), patient-reported outcomes and digital measures (see outcome measures).

Detailed motor assessments are included in the following cohorts: B (older healthy controls), C (SCD/MCI with suspicion of incipient neurocognitive disorder) and E (parkinsonian disorders).

CEREBROSPINAL FLUID (CSF) AND BLOOD SAMPLING AND ANALYZES Lumbar CSF samples will be collected according to a standardized protocol and will follow the principles of the Alzheimer's Association Flow Chart for CSF biomarkers. In short, lumbar puncture will be done between 9-12 am. 20-30 ml of CSF will be collected in Low Binding polypropylene tubes, which are stored on ice for 5-20 min until the CSF samples will be centrifuged (2000g, +4°C, 10 min). Thereafter, the CSF will be aliquoted in ca 1 ml portions into Low Binding polypropylene tubes followed by storage at -80°C until batch analyses.

Plasma collection will be done at the same visit as the lumbar puncture. Blood will be drawn into tubes containing either EDTA (5 x 6 ml tubes) or Lithium heparin (3 x 3 ml tubes) as anticoagulant. After centrifugation (2000g, +4°C, 10 min), plasma samples will be aliquoted into polypropylene tubes and stored at -80°C pending biochemical analyses. Further, EDTA-blood (2 x 6 ml) will also be obtained for genetic DNA analyses.

MAGNETIC RESONANCE IMAGING 3 Tesla MRI (Siemens Prisma) will be done in all study cohorts. A wide variety of magnetic resonance imaging (MRI) techniques will be used to study regional brain volume (three-dimensional magnetization-prepared rapid acquisition with gradient echo (3D MPRAGE)), metabolism (MR spectroscopy (MRS)), structural and functional connectivity of different brain regions (diffusion tensor imaging (DTI) and functional MRI (fMRI)), regional blood flow (arterial spin labeling (ASL)), iron deposition (susceptibility-weighted imaging (SWI)) and the presence of small vessel disease (MPRAGE, SWI and fluid-attenuated inversion recovery (FLAIR)). The protocol will take approximately 60 min to perform. No contrast-enhancing agent will be used.

PET IMAGING

Tau PET. PET imaging of tau aggregates will be done in all the included cohorts at baseline. In the present study, Tau PET imaging will be performed using 18F-RO6958948 developed by Hoffmann-La Roche that will provide the precursor for this PET ligand. This tau PET imaging agent has been shown to accurately detect tau pathology in cases with AD when compared to controls. We will perform a 20-30 min PET scan approximately 60 min post intravenous injection of 18F-RO6958948. The impact of the investigation on clinical diagnostic accuarcy and patient care will be investigated. 18F-RO6958948 has not yet been approved for use in clinical routine practice in Sweden, and can only be used in research studies, such as the present study.

Amyloid PET. PET imaging of Aβ aggregates (including 18F-flutemetamol PET) has been approved for use in clinical routine practice in Sweden. In the present study, 18F-flutemetamol PET will be done in non-demented cases only. In the cases with dementia CSF Aβ will be enough to determine the presence or absence of brain amyloid pathology. However, in the cognitively healthy cases and in the patients with SCD or MCI we are interested in following the spread of amyloid pathology throughout the brain during the preclinical stages of AD and the spatial relationship to tau pathology. Therefore, Amyloid PET will be done according to clinical routine procedures in addition to CSF Aβ measurements in these groups. In the present study Amyloid PET will be performed using 18F-flutemetamol. GE Healthcare will provide the precursor for 18F-flutemetamol. A 20 min scan will be performed between 90-110 min post injection of 18F-flutemetamol.

FDOPA PET FDOPA PET is often used as part of clinical routine examinations of patients with parkinsonism to confirm the diagnosis. Here DaTSCAN will be done according to clinical routine procedures in cases with PD, PDD, DLB, MSA, PSP and CBD to confirm the clinical diagnosis if it has not been done in clinical routine praxis within one year from the baseline visit.

ELIGIBILITY:
COHORT A: Cognitively healthy younger individuals (40-65 years of age) INCLUSION CRITERIA

* Age 40-65 years
* Absence of cognitive symptoms as assessed by a physician with special interest in cognitive disorders.
* MMSE score 27-30 at screening visit.
* Do not fulfill the criteria for MCI or any dementia according to DSM-V.
* Speaks and understands Swedish to the extent that an interpreter is not necessary for the patient to fully understand the study information and cognitive tests.

EXCLUSION CRITERIA

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Significant neurological or psychiatric illness.
* Refusing lumbar puncture, MRI or PET.

COHORT B: Cognitively healthy elderly individuals (66-100 years of age) INCLUSION CRITERIA

* Age 66-100 years
* Absence of cognitive symptoms as assessed by a physician with special interest in cognitive disorders.
* MMSE score 26-30 at screening visit.
* Do not fulfill the criteria for MCI or any dementia according to DSM-V.
* Speaks and understands Swedish to the extent that an interpreter is not necessary for the patient to fully understand the study information and cognitive tests.

EXCLUSION CRITERIA

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Significant neurological or psychiatric illness.
* Refusing lumbar puncture, MRI or PET.

COHORT C: Subjective cognitive decline and mild cognitive impairment INCLUSION CRITERIA

* Age 40-100 years.
* Referred to the memory clinics due to cognitive symptoms experienced by the patient and/or informant. These symptoms do not have to be memory complaints, but could also be executive, visuospatial, language, praxis, psychomotor or social cognitive complaints.
* MMSE score of 24 - 30 points.
* Do not fulfill the criteria for any dementia (major neurocognitive disorder) according to DSM-V.
* The medical doctor (after clinical assessments, cognitive testing, CSF analyses and structural brain imaging) believes the cognitive complaints are caused by an incipient neurocognitive disorder of any sort. This is defined as any case fulfilling the criteria above (i.e. both SCD and MCI) with an abnormal CSF Aβ42/40 ratio, which is strongly associated with brain Aβ pathology and prodromal Alzheimer's disease. Further, cases with MCI (=minor neurocognitive impairment) due to either Parkinson's disease, Lewy body disease, vascular neurocognitive disorder or frontotemporal dementia (please see Appendix below for clinical criteria and references) can also be included.
* Speaks and understands Swedish to the extent that an interpreter is not necessary for the patient to fully understand the study information and cognitive tests.

EXCLUSION CRITERIA

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Refusing lumbar puncture, MRI or PET.

COHORT D: Dementia due to Alzheimer's disease INCLUSION CRITERIA

* Age 40-100 years.
* Referred to the memory clinics due to cognitive symptoms experienced by the patient and/or informant. These symptoms do not have to be memory complaints, but could also be executive, visuospatial, language, praxis or psychomotor complaints.
* MMSE score of 12-26 points.
* Fulfill the criteria for dementia (major neurocognitive disorder) due to Alzheimer's disease (DSM-V).
* Speaks and understands Swedish to the extent that an interpreter was not necessary for the patient to fully understand the study information and cognitive tests.

EXCLUSION CRITERIA

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Refusing lumbar puncture, MRI or PET.

COHORT E: Other dementias INCLUSION CRITERIA

* Age 40-100 years.
* Fulfill the criteria for dementia (major neurocognitive disorder) due to FTD, PDD, DLB or subcortical VaD alternatively the criteria for PD, PSP, MSA or CBS.
* Speaks and understands Swedish to the extent that an interpreter was not necessary for the patient to fully understand the study information and cognitive tests.

EXCLUSION CRITERIA

* Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
* Current significant alcohol or substance misuse.
* Refusing lumbar puncture, MRI or PET.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1505 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical diagnosis | Clinical diagnosis at last 1 day visit
  Clinical diagnosis according to consensus group decision blinded to the diagnostic test
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 2-8 years after baseline.
  Change in CDR-SB

SECONDARY OUTCOMES:
Rate of cognitive decline as measured by MMSE. | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 2-8 years after baseline.
  Mini Mental State Examination (MMSE)
Rate of cognitive decline as measured in ADL-function. | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 2-8 years after baseline.
  ADL function will be determined using the Functional Assessment Questionnaire (FAQ) and The Amsterdam ADL scale
Rate of volume change of structural MRI measures and amyloid PET | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 2-8 years after baseline.
Rates of change on cerebrospinal fluid AD biomarkers | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for approximately 2-8 years after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Hansson, MD, Professor, Principal Investigator — Skåne University Hospital, and Lund University
Locations (2):
- Sweden (2):
  - Memory Clinic, Hospital of Ängelholm, Ängelholm
  - Memory Clinic, Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cullen N, Janelidze S, Palmqvist S, Stomrud E, Mattsson-Carlgren N, Hansson O; Alzheimer's Disease Neuroimaging Initiative. Association of CSF Abeta38 Levels With Risk of Alzheimer Disease-Related Decline. Neurology. 2022 Mar 1;98(9):e958-e967. doi: 10.1212/WNL.0000000000013228. Epub 2021 Dec 22. PMID 34937781